CLINICAL TRIAL: NCT03902678
Title: Role of Endoscopic Ultrasound Guided Fine Needle Aspiration of Portal Vein Thrombus in the Diagnosis and Staging of Hepatocellular Carcinoma
Brief Title: Role of EUS Guided FNA of Portal Vein Thrombus in the Diagnosis and Staging of Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MD /17.06.69
Record Dates: First submitted 2019-01-26; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Portal Vein Thrombosis
Keywords: EUS; FNA; PVT

STUDY DESIGN:
Intervention Model Description: Use of histopathology obtained from endoscopic ultrasound -fine needle aspiration of portal vein thrombus for identification of malignant thrombus which did not fulfill criteria of malignancy by abdominal ultrasound and triphasic abdominal CT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EUS - FNA for benign PVT by imaging (Experimental): Intervention: Procedure/Surgery: EUS guided fine needle aspiration of portal vein thrombus
  Interventions: Procedure: EUS guided fine needle aspiration of portal vein thrombus

INTERVENTIONS:
Procedure: EUS guided fine needle aspiration of portal vein thrombus — endoscopic ultrasound guided fine needle aspiration of portal vein thrombus which did not fulfill criteria of malignancy by imaging technique

SUMMARY:
Since not every portal vein thrombus (PVT) in a patient with hepatocellular carcinoma (HCC) is a tumor thrombus, since the nature of the thrombus will ultimately determine the course of treatment, and since PVT may be even the initial sign of an undetected HCC, every effort should be made to distinguish between a tumor and a non-tumor PVT. In addition, malignant PVT does not always demonstrate neovascularity and/or enhancement, which makes fine needle aspiration (FNA) necessary in order to characterize the nature of the PVT.

Sampling of portal vein thrombus with trans-abdominal ultrasound guidance may lead to erroneous results because of inadvertent inclusion of normal hepatocytes or associated liver masses. Further, potential adverse events of trans-abdominal portal vein sampling include serious biliary and/or vascular injury.

In contrast to the percutaneous approach, Endoscopic ultrasound (EUS) provides a unique view and access to the main portal vein. From the duodenal bulb and second part of the duodenum, the portal vein can be visualized from the confluence of the splenic and superior mesenteric veins into the porta hepatis. Periportal collateral vessels or cavernous transformation of the portal vein, which commonly are associated with portal vein thrombosis, are also easily and reliably detected by EUS instruments with color Doppler US capability.

With a linear-array echo-endoscope, the portal vein can be punctured easily with a fine needle under direct visualization, while avoiding the adjacent hepatic artery, bile duct, and collateral vessels (if present). Because the approach is not trans-hepatic, it eliminates any need to avoid the primary tumor and any possibility of contaminating the specimen with hepatocytes, as can occur if the needle tracks through the liver parenchyma. Thus, the rate of false-positive diagnoses is likely to be lower with the EUS compared with the percutaneous approach

DETAILED DESCRIPTION:
This is a pilot study that include 30 patients with liver cirrhosis and portal vein thrombus which don't fulfill the criteria of malignancy by imaging technique. The patients involved in the study were and will be admitted to Specialized Medical Hospital, Mansoura University Hospitals.

Study end-points:

• 24 months from the start of the research (cases will be collected over 18 months).

Methods:

Patients will be included in this study will be subjected to the following:

І. The study will be explained to all participants in the study, and an informed written consent will be obtained from them before starting the study.

ІІ. Medical history:

Detailed history was taken with stress on:

* Signs of cachexia (unintentional weight loss, progressive muscle wasting, and a loss of appetite)
* Low grade fever
* Recent onset fatigue
* Abdominal pain
* Dyspepsia
* Hematemesis and melena
* Back ache

ІІІ. Full clinical examination with special stress on:

* Vital signs including: pulse, arterial blood pressure, temperature, respiratory rate.
* Abdominal Lumps and/or tenderness

IV. Laboratory investigations:

Complete blood count, International Normalized Ratio, Liver enzymes, Serum albumin, Serum bilirubin and Serum creatinine.

V. Radiology: Abdominal ultrasound for initial assessment, Abdominal CT (Contrast Enhanced) (Number of HCC nodules if present, diameter of largest HCC nodule in centimeters, nature of PVT, presence of abdominal metastases if present ), Non contrast CT chest to exclude pulmonary metastasis, Bone survey for indicated or complaining cases.

VI. EUS-FNA:

EUS-FNA will be performed in standard fashion. Under EUS guidance, the main, left and right portal veins will be identified. After verifying flow signal by Doppler, a 25-gauge EUS-FNA needle will be advanced from the duodenal bulb or second part of the duodenum into the portal vein, 1-2 passes through portal vein thrombus will be taken to ensure adequate cellularity for histopathology. The puncture site will be monitored under EUS for complications.

Study outcomes:

Histopathology of biopsies taken from bland portal vein thrombus which diagnosed by triphasic CT abdomen to evaluate the possibility of malignant PVT that was not discovered by imaging technique (Abdominal ultrasound and triphasic abdominal CT ).

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver cirrhosis and PVT which don't fulfill criteria of malignancy by triphasic CT abdomen defined as, (neovascularity of thrombus, arterial enhancement with rapid washout, direct invasion by adjacent hepatic mass and diameter of thrombus more than 23 mm), either :
* With or without hepatic mass
* Undergone local treatment or surgical treatment following a diagnosis of HCC and develop PVT during their follow up.

Exclusion Criteria:

* Uncooperative or excessively apprehensive patient
* Anticoagulation treatment or non-substituted coagulopathy (International Normalized Ratio ≥ 1.5, Platelet count ≤ 50.000 cells/mm3, heparin administration at therapeutic doses).
* Inhibition of platelet aggregation by clopidogrel and other thienopyridines.
* Contraindications of sedation (Uncontrolled Diabetes Mellitus, Uncontrolled Thyroid Disorders, Pregnancy, Respiratory Embarrassment, Reactional Drugs like Antidepressants and Anti-anxiety Agents).
* Patients fulfilling criteria of malignancy by triphasic CT on abdomen.
* Extra hepatic metastasis of HCC.
* Child-Pugh classification stage C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-11 (Actual); Primary Completion 2019-05-11 (Estimated); Study Completion 2019-07-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with bland portal vein thrombosis diagnosed by triphasic abdominal CT who are proven to have malignant cells by histopathology obtained via EUS-guided FNA | 3 days up to 2 weeks
  Histopathology of biopsies taken from bland portal vein thrombus which diagnosed by triphasic CT abdomen to evaluate the possibility of malignant PVT that was not discovered by imaging technique (Abdominal ultrasound and triphasic abdominal CT )
Percentage of patients with portal vein thrombosis who underwent EUS guided FNA and had complications as a result of the invasive maneuver | 2 days
  assessment of safety of the procedure ( The patients admitted and the new ones will be admitted to specialized medical hospital for 24 h after the procedure to exclude the possibility of bleeding at puncture site, risk of biliary peritonitis, and extravasation from the site of the thrombus.

CONTACTS AND LOCATIONS:
Overall Officials: Magdy H. Atwa, Professor, Study Chair — Faculty of Medicine, Mansoura University
Locations (1):
- specialized medical hospital, Mansourah University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catalano OA, Choy G, Zhu A, Hahn PF, Sahani DV. Differentiation of malignant thrombus from bland thrombus of the portal vein in patients with hepatocellular carcinoma: application of diffusion-weighted MR imaging. Radiology. 2010 Jan;254(1):154-62. doi: 10.1148/radiol.09090304. PMID 20032150
- [Background] Handa P, Crowther M, Douketis JD. Portal vein thrombosis: a clinician-oriented and practical review. Clin Appl Thromb Hemost. 2014 Jul;20(5):498-506. doi: 10.1177/1076029612473515. Epub 2013 Jan 29. PMID 23364162
- [Background] Lai R, Stephens V, Bardales R. Diagnosis and staging of hepatocellular carcinoma by EUS-FNA of a portal vein thrombus. Gastrointest Endosc. 2004 Apr;59(4):574-7. doi: 10.1016/s0016-5107(04)00007-0. No abstract available. PMID 15044903
- [Background] Tarantino L, Ambrosino P, Di Minno MN. Contrast-enhanced ultrasound in differentiating malignant from benign portal vein thrombosis in hepatocellular carcinoma. World J Gastroenterol. 2015 Aug 28;21(32):9457-60. doi: 10.3748/wjg.v21.i32.9457. PMID 26327753
- [Background] ASGE Technology Committee; Trikudanathan G, Pannala R, Bhutani MS, Melson J, Navaneethan U, Parsi MA, Thosani N, Trindade AJ, Watson RR, Maple JT. EUS-guided portal vein interventions. Gastrointest Endosc. 2017 May;85(5):883-888. doi: 10.1016/j.gie.2017.02.019. Epub 2017 Mar 18. No abstract available. PMID 28320514
- [Background] Viechtbauer W, Smits L, Kotz D, Bude L, Spigt M, Serroyen J, Crutzen R. A simple formula for the calculation of sample size in pilot studies. J Clin Epidemiol. 2015 Nov;68(11):1375-9. doi: 10.1016/j.jclinepi.2015.04.014. Epub 2015 Jun 6. PMID 26146089
- [Result] Kayar Y, Turkdogan KA, Baysal B, Unver N, Danalioglu A, Senturk H. EUS-guided FNA of a portal vein thrombus in hepatocellular carcinoma. Pan Afr Med J. 2015 Jun 3;21:86. doi: 10.11604/pamj.2015.21.86.6991. eCollection 2015. PMID 26491529
- [Result] Michael H, Lenza C, Gupta M, Katz DS. Endoscopic Ultrasound -guided Fine-Needle Aspiration of a Portal Vein Thrombus to Aid in the Diagnosis and Staging of Hepatocellular Carcinoma. Gastroenterol Hepatol (N Y). 2011 Feb;7(2):124-9. No abstract available. PMID 21475421
- [Result] Rustagi T, Gleeson FC, Chari ST, Abu Dayyeh BK, Farnell MB, Iyer PG, Kendrick ML, Pearson RK, Petersen BT, Rajan E, Topazian MD, Truty MJ, Vege SS, Wang KK, Levy MJ. Remote malignant intravascular thrombi: EUS-guided FNA diagnosis and impact on cancer staging. Gastrointest Endosc. 2017 Jul;86(1):150-155. doi: 10.1016/j.gie.2016.10.025. Epub 2016 Oct 20. PMID 27773725
- See also: paper proved that benign portal vein thrombus by triphasic CT may be truly malignant by the histopathology but the researchers here used different inclusion and exclusion criteria. They obtained samples from cirrhotic patients only — http://www.pulmonarychronicles.com/index.php/pulmonarychronicles/article/view/496

DOCUMENTS (1):
  • Study Protocol (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT03902678/Prot_000.pdf